CLINICAL TRIAL: NCT03757143
Title: Skin Antisepsis With Chlorhexidine-Alcohol Versus Povidone Iodine-Alcohol, Combined or Not With Use of a Bundle of New Devices, for Prevention of Intravascular-catheter Colonization and Catheter Failure: An Open Label, Single Center, Randomized Controlled, Two-by-two Factorial Trial
Brief Title: Chlorhexidine-Alcohol Versus Povidone Iodine-Alcohol, Combined or Not With Use of a Bundle of New Devices, for Prevention of Intravascular-catheter Colonization and Catheter Failure
Acronym: CLEAN3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CLEAN3
Record Dates: First submitted 2018-11-27; First posted 2018-11-28 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Intravascular-catheter Colonization; Catheter Failure
Keywords: Skin antisepsis; Chlorhexidine; Povidone Iodine; Intravascular-catheter colonization; Catheter failure; Bundle of new devices
MeSH Terms: interventions — Povidone-Iodine; Ethanol; Chlorhexidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PVI et Insyte (Active Comparator): Groupe A: (1) 5% (w/v) PVI-69% (v/v) ethanol (Bétadine alcoolique™, MEDA Pharma SAS); (2) InsyteTM AutoguardTM BC Winged, BD
  Interventions: Drug: Povidone-Iodine-Alcohol; Device: Insyte Autoguard BC Winged
- CHG et Insyte (Experimental): Groupe B: (1) 2% (w/v) CHG-70% (v/v) isopropanol (ChloraPrep™, CareFusion); (2) InsyteTM AutoguardTM BC Winged, BD
  Interventions: Drug: Chlorhexidine-Alcohol; Device: Insyte Autoguard BC Winged
- PVI et Nexiva (Experimental): Groupe C: (1) 5% (w/v) PVI-69% (v/v) ethanol (Bétadine alcoolique™, MEDA Pharma SAS); (2) NexivaTM single port catheter, MaxZeroTM needleless connector, , PureHub™ Desinfecting Caps, PosiflushTM prefilled saline syringes, all from BD
  Interventions: Drug: Povidone-Iodine-Alcohol; Device: Nexiva single port catheter, MaxZero needless connector, PureHub Deinfecting Caps and Posiflush prefilled saline syringes
- CHG et Nexiva (Experimental): Groupe D: (1) 2% (w/v) CHG-70% (v/v) isopropanol (ChloraPrep™, CareFusion); (2) NexivaTM single port catheter, MaxZeroTM needleless connector, PureHub™ Desinfecting Caps, PosiflushTM prefilled saline syringes, all from BD
  Interventions: Drug: Chlorhexidine-Alcohol; Device: Nexiva single port catheter, MaxZero needless connector, PureHub Deinfecting Caps and Posiflush prefilled saline syringes

INTERVENTIONS:
Drug: Povidone-Iodine-Alcohol — Povidone-Iodine-Alcohol will be used to disinfect the skin
  Arms: PVI et Insyte; PVI et Nexiva
Drug: Chlorhexidine-Alcohol — Chlorhexidine-Alcohol will be used to disinfect the skin
  Arms: CHG et Insyte; CHG et Nexiva
Device: Insyte Autoguard BC Winged — Pose of Insyte Autoguard BC Winged
  Arms: CHG et Insyte; PVI et Insyte
Device: Nexiva single port catheter, MaxZero needless connector, PureHub Deinfecting Caps and Posiflush prefilled saline syringes — Pose of Nexiva single port catheter
  Arms: CHG et Nexiva; PVI et Nexiva

SUMMARY:
Short peripheral intravenous catheters (PVC) are the most frequently used invasive medical devices in hospitals. Unfortunately, PVCs often fail before the end of treatment due to the occurrence of complications, which can be mechanical, vascular or infectious. Complications lead to infusion failure and device replacement, which results in interrupted therapy, pain associated with resiting and increased health care costs for resources and staff time. Catheter related bloodstream infections (CR-BSIs) prolong hospitalization and increase treatment costs and mortality.

Prevention of these complications is based on the respect of hygiene rules and the use of bio-compatible catheters. The choice of the antiseptic solution for skin disinfection is key. Similarly, the use of new technologies such as catheters designed to minimize blood exposure, zero-reflux needleless-connectors, disinfecting caps, and flushing PVCs before and after each medication administration to maintain catheter patency are of theoretical interest, but little scientific data support their use in routine.

The primary objectives of this study are, first, to demonstrate that skin preparation with 2% chlorhexidine (CHG)-70% isopropanol decreases the risk of PVC colonization compared to skin preparation with 5% povidone iodine (PVI)-69% ethanol. Second, to demonstrate that use of a bundle of technologies including a new PVC, zero-reflux needless-connectors, disinfecting caps, and single-use prefilled flush syringes extends the time between catheter insertion and catheter failure.

The secondary objectives are to compare between the four study group incidence of phlebitis, accidental catheter removal, infiltration, catheter occlusion, CR-BSI, local infection, all-cause bloodstream infections, catheter colonization, duration of catheter remaining in place without complication, length of hospital stay, safety and patient satisfaction.

The CLEAN 3 study is an open-label, single centre, investigator-initiated, randomised, four-parallel group, two-by-two factorial trial. Patients requiring PVC for an expected 48 h will be randomised in one of four groups according to skin disinfection method and type of devices used. Randomization will be carried out through a secure web-based randomization system. Inclusions are expected to begin in January 2019 and continue until July 2019, once the number of catheters required has been reached.

Patients will be enrolled at the Emergency department of the Poitiers University Hospital before being hospitalised in one of five wards (neurology, neurology, pneumology, internal medicine and downstream emergency unit).

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥ 18 years) patients,
* Having clinical indication for placement of a single PVC for at least 48 hours (no minimum port access during the study duration),
* Willing and able to provide informed consent.

Exclusion Criteria:

* Known allergies to CHG, PVI, isopropanol or ethanol,
* Participation to another clinical trial aimed at reducing PVC complications,
* Suspicion of bloodstream infection at catheter insertion,
* Skin injury a catheter insertion site increasing the risk of catheter infection,
* PVC inserted extremely urgently, making it impossible to comply with the protocol,
* Intravascular catheter in place within the last 2 days, or within the last 2 weeks and with local signs of catheter complication,
* Difficult catheter insertion suspected (obesity, known IV drug users, non-visible venous network after placement of a tourniquet...),
* Patients already enrolled in this study,
* Terminal or moribund patient not expected to live more than one week,
* Patients not benefiting from a Social Security scheme or not benefiting from it through a third party,
* Persons benefiting from enhanced protection, namely minors, persons deprived of their liberty by a judicial or administrative decision, adults under legal protection.
* Pregnant or breastfeeding women
* Women at age to procreate and not using effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-27 (Actual)

PRIMARY OUTCOMES:
Incidence of catheter-related infectious complications | 8 days
  Incidence of catheter-related infectious complications, and include catheter colonisation, local infection and CR-BSI
Time between catheter insertion and catheter failure | 8 days
  Time between catheter insertion and catheter failure: defined as any premature removal of PVC before end of treatment, other than for routine replacement, and includes phlebitis, infiltration, occlusion, accidental catheter removal, local infection and CR-BSI whichever occurred first

SECONDARY OUTCOMES:
Number of phlebitis | 8 days
  Number of phlebitis defined as two or more of the following present simultaneously: (1) patient-reported pain or tenderness (on questioning, then palpation by the research nurse) with a severity of two or more on a ten-point scale; (2) erythema extending at least 1 cm from the insertion site; (3) swelling, extending at least 1 cm from the insertion site; (4) purulent discharge; or (5) palpable venous cord beyond the intravenous catheter tip
Number of accidental catheter removal | 8 days
Number of infiltration | 8 days
  Number of infiltration, defined as the infusion of non-blistering drug leaking through the normal vascular channel and resulting in the swelling of tissue peripheral to the puncture site
Number of catheter occlusion | 8 days
  Number of catheter occlusion defined as the inability of the catheter to flush (not able to intravenously inject 1ml of normal saline within 30 s)
Number of CR-BSI | 8 days
  Number of CR-BSI, defined as (1) at least one positive blood culture from a peripheral vein and (2) clinical signs of infection (ie, fever [body temperature >38°5], hypothermia [body temperature <36°5], chills, or hypotension [Systolic blood pressure <90 mm Hg]) and (3) no other apparent source for the bloodstream infection except the PVC (in situ within 48 h of the bloodstream infection); and (4) a colonized intravenous catheter tip culture with the same organism (same species) as identified in the blood. For commensal micro-organisms (coagulase-negative staphylococci, Corynebacterium spp. [except C. jeikeium], Lactobacillus spp., Bacillus spp. and Propionibacterium spp., or viridans group Streptococcus isolates and C. perfringens) at least two positive blood cultures will be required.
Number of local infection | 8 days
  Number of local infection, defined as organisms grown from purulent discharge with no evidence of associated bloodstream infection
Number of all-cause bloodstream infections | 8 days
  Number of all-cause bloodstream infections, defined as any positive blood culture drawn from a peripheral vein while intravenous catheter in situ or for 48 h after removal. For commensal micro-organisms (coagulase-negative staphylococci, Corynebacterium spp. [except C. jeikeium], Lactobacillus spp., Bacillus spp. and Propionibacterium spp., or viridans group Streptococcus isolates and C. perfringens) at least two positive blood cultures will be required
Number of catheter colonization | 8 days
  Number of catheter colonization defined as the culture of intravascular catheter tip showing at least 1000 colony-forming units per ml (cfu/ml).
Number of pathogens involved in catheter colonization, local infections, CR-BSI and all-cause bloodstream infections | 8 days
Number of days the catheter remaining in place without complication | 8 days
Length of Hospital stay censored at day 28 | 28 days
Incidence of local and systemic side effects possibly linked to antiseptic use | 8 days
Patient's evaluation of the pain at the insertion of the catheter using visual analogue scale (VAS) | 8 days
  Visual analogue scale is increased from 0 to 10, 0 is the better outcome (no pain) and 10 is the worse outcome
Patient's satisfaction at catheter removal using visual analogue scale (VAS) | 8 days
  Visual analogue scale is increased from 0 to 10, 0 is the worse outcome (no satisfaction) and 10 is the better outcome
Evaluation impact of venous line on patients' mobility at catheter removal using visual analogue scale | 8 days
  Visual analogue scale is increased from 0 to 10, 0 is the better outcome (no impact of patients'mobility) and 10 is the worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Poitiers, Poitiers, France

REFERENCES:
- [Derived] Maunoury F, Drugeon B, Boisson M, Marjanovic N, Couvreur R, Mimoz O, Guenezan J; CLEAN-3 Study. Cost-effectiveness analysis of bundled innovative devices versus standard approach in the prevention of unscheduled peripheral venous catheters removal due to complications in France. PLoS One. 2022 Jun 14;17(6):e0269750. doi: 10.1371/journal.pone.0269750. eCollection 2022. PMID 35700207
- [Derived] Guenezan J, Marjanovic N, Drugeon B, Neill RO, Liuu E, Roblot F, Palazzo P, Bironneau V, Prevost F, Paul J, Pichon M, Boisson M, Frasca D, Mimoz O; CLEAN-3 trial investigators. Chlorhexidine plus alcohol versus povidone iodine plus alcohol, combined or not with innovative devices, for prevention of short-term peripheral venous catheter infection and failure (CLEAN 3 study): an investigator-initiated, open-label, single centre, randomised-controlled, two-by-two factorial trial. Lancet Infect Dis. 2021 Jul;21(7):1038-1048. doi: 10.1016/S1473-3099(20)30738-6. Epub 2021 Feb 1. PMID 33539734
- [Derived] Guenezan J, Drugeon B, O'Neill R, Caillaud D, Senamaud C, Pouzet C, Seguin S, Frasca D, Mimoz O. Skin antisepsis with chlorhexidine-alcohol versus povidone iodine-alcohol, combined or not with use of a bundle of new devices, for prevention of short-term peripheral venous catheter-related infectious complications and catheter failure: an open-label, single-centre, randomised, four-parallel group, two-by-two factorial trial: CLEAN 3 protocol study. BMJ Open. 2019 Apr 2;9(4):e028549. doi: 10.1136/bmjopen-2018-028549. PMID 30944142